CLINICAL TRIAL: NCT05640752
Title: Optimal Evaluation of Stable Chest Pain to Reduce Unnecessary Utilization of Cardiac Imaging Testing
Brief Title: Optimal Evaluation to Reduce Cardiovascular Imaging Testing
Acronym: OPERATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhou Jia, Principal Investigator, Tianjin Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2022KY-024-01; 62206197 (Other Grant/Funding Number: National Natural Science Foundation of China); TJWJ2022QN067 (Other Grant/Funding Number: Tianjin Health Research Project); 21JCYBJC00820 (Other Grant/Funding Number: Applied and Basic Research by Multi-input Foundation of Tianjin)
Record Dates: First submitted 2022-11-27; First posted 2022-12-07 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Coronary Syndrome
Keywords: Stable Chest Pain; Pretest Probability; Coronary Computed Tomography Angiography; Diagnostic Strategy; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESC strategy (Experimental): ESC-PTP is calculated using age, sex and type of chest pain according to 2019 ESC guideline for the diagnosis and management of CCS and RF-CL is calculated using age, sex, type of chest pain, hypertension, dyslipidemia, diabetes, smoking and family history of CAD based on the publication of Winther et al., respectively. According to ESC strategy, subjects with ESC-PTP ≤5% are classified into low risk group and ones with ESC-PTP ≥15% are classified into high risk group. For subjects with ESC-PTP of 5%-15%, ones with RF-CL ≥15% are classified into high risk group and ones with RF-CL <15% are classified into low risk group. CCTA should be referred for a subject in high risk group. Subjects determined to be at low risk will be referred to optimal medication treatment with no immediate CCTA.
  Interventions: Diagnostic Test: 2019 ESC guideline-determined diagnostic strategy
- NICE strategy (Experimental): According to NICE strategy, subjects with nonanginal chest pain and normal ECG are classified into low risk group and ones with typical and atypical angina or nonanginal chest pain with abnormal ECG are classified into high risk group. CCTA should be referred for a subject in high risk group. Subjects determined to be at low risk will be referred to optimal medication treatment with no immediate CCTA.
  Interventions: Diagnostic Test: 2016 NICE guideline-determined diagnostic strategy

INTERVENTIONS:
Diagnostic Test: 2019 ESC guideline-determined diagnostic strategy — ESC-PTP is calculated using age, sex and type of chest pain according to 2019 ESC guideline for the diagnosis and management of CCS and RF-CL is calculated using age, sex, type of chest pain, hypertension, dyslipidemia, diabetes, smoking and family history of CAD based on the publication of Winther et al., respectively. According to ESC strategy, subjects with ESC-PTP ≤5% are classified into low risk group and ones with ESC-PTP ≥15% are classified into high risk group. For subjects with ESC-PTP of 5%-15%, ones with RF-CL ≥15% are classified into high risk group and ones with RF-CL <15% are classified into low risk group. CCTA should be referred for a subject in high risk group. Subjects determined to be at low risk will be referred to optimal medication treatment with no immediate CCTA.
  Arms: ESC strategy
Diagnostic Test: 2016 NICE guideline-determined diagnostic strategy — For subjects assigned to NICE strategy, ones with nonanginal chest pain and normal ECG were classified into low risk group and ones with typical and atypical angina or nonanginal chest pain with abnormal ECG were classified into high risk group. Subjects determined to be at low risk will be referred to optimal medication treatment with no immediate CCTA.
  Arms: NICE strategy

SUMMARY:
In daily clinical routine, the evaluation of new-onset and stable chest pain (SCP) suggestive of chronic coronary syndrome (CCS) remains a challenge for physicians. Although coronary computed tomography angiography (CCTA) seems to be the first-line cardiac imaging testing (CIT) according to the recommendations from current guidelines, the optimal diagnostic strategy to identify low risk patients who may derive minimal benefit from further CIT is the cornerstone of clinical management for SCP. Recently, different diagnostic strategies were provided to effectively defer unnecessary CIT, but few studies have prospectively determined the actual effect of applying these strategies in clinical practice. Therefore, the OPERATE study was designed to compare the effectiveness and safety of two proposed diagnostic strategies in identification of low risk individual who may derive minimal benefit from CCTA among patients with SCP suggestive of CCS in a pragmatic randomized controlled trial (RCT).

DETAILED DESCRIPTION:
OPERATE trial was an investigator-initiated, multicenter, prospective, CCTA-based, 2-arm 1:1 parallel-group, double-blind and pragmatic RCT planned to include 800 subjects with SCP suggestive of CCS. Subjects were assigned randomly to two groups: 1) 2016 National Institutes for Clinical Excellence guidelines-determined diagnostic strategy (NICE strategy) and 2) 2019 European Society of Cardiology guidelines-determined diagnostic strategy (ESC strategy) The primary objective of OPERATE trial is to compare the rates of CCTA without obstructive CAD according to NICE and ESC strategy. The key secondary objective is to assess whether the two strategies have no significant difference in terms of major adverse cardiac events (MACE). The investigators hypothesize that when comparing with NICE strategy, ESC strategy which sequentially incorporated the ESC-PTP model with RF-CL model will decrease the probability of CCTA without obstructive CAD but not at the expense of safety and cost over a follow-up period of 1 year.

ELIGIBILITY:
Inclusion criteria

1. SCP or equivalenta suggestive of CCS and clinically stability
2. No history of CAD (prior myocardial infarction, CR or any CAD documented by previous CIT)
3. Age ≥30 years
4. Willing and able to provide informed consent

Exclusion criteria

1. Prior CIT within 1 year prior to randomization
2. Clinically instability (e.g. cardiogenic shock, ACS, severe arrhythmias or NYHA III or IV heart failure)
3. Non-sinus rhythm
4. Concomitant participation in another clinical trial
5. Complex structural heart disease
6. Non-cardiac illness with life expectancy < 2 years
7. Allergy to iodinated contrast agent
8. Estimated glomerular filtration rate<60 ml/min/1.73m2 within 90 days
9. Body mass index >35kg/m2
10. Expressing a clear preference for undergoing CIT or not
11. Pregnancy

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
CCTA without obstructive CAD | Through the initial management, an average of 2-5 days
  The summary of nonobstructive CAD, no sign of CAD and nondiagnostic result detected by CCTA according to each strategy

SECONDARY OUTCOMES:
MACE | 1 year
  All-cause death, myocardial infarction and hospitalization due to unstable angina.
All-cause death | 1 year
  Any death.
Myocardial infarction | 1 year
  Myocardial infarction was defined and classified as spontaneous or coronary procedure-related MI according to the Fourth Universal Definition of Myocardial Infarction.
Hospitalization due to unstable angina | 1 year
  An hospitalization event in which the final diagnosis was myocardial ischemia.
Exposure to radiation | 1 year
  All exposure to radiation related to CIT and other cardiovascular procedures.
Procedural complications | 1 year
  All procedural complications related to CIT and other cardiovascular procedures.
Cumulative proportion of patients receiving other CITs | 1 year
Cumulative proportion of patients receiving CR | 1 year
Cumulative proportion of patients who had alteration in OMT based on results of CCTA | Thtough the initial management, an average of 2-5 days
Proportion of normal CCTA | Through the initial management, an average of 2-5 days
Proportion of necessary CCTA | Through the initial management, an average of 2-5 days

OTHER OUTCOMES:
The health-related quality of life assessment (SAQ) | 1 year
  Seattle Angina Questionnaire
The health-related quality of life assessment (EQ-5D) | 1 year
  Visual-analogue scale of the European Quality of Life-5 Dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, MD, Principal Investigator — Tianjin Chest Hospital
Locations (4):
- China (4):
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Hebei Petrochina Central Hospital, Lanfang, Hebei
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou J, Xin T, Tan Y, Pang J, Chen T, Wang H, Zhao J, Liu C, Xie C, Wang M, Wang C, Liu Y, Zhang J, Liu Y, Shanfu C, Li C, Cong H. Comparison of two diagnostic strategies for patients with stable chest pain suggestive of chronic coronary syndrome: rationale and design of the double-blind, pragmatic, randomized and controlled OPERATE Trial. BMC Cardiovasc Disord. 2023 Aug 23;23(1):416. doi: 10.1186/s12872-023-03424-3. PMID 37612631